CLINICAL TRIAL: NCT03356236
Title: A Multicenter, Prospective Cohort Study Investigating Huaier Granule for Prevention of Recurrence and Metastasis of Hepatocarcinoma Following Local Ablation
Brief Title: Huaier Granule for Prevention of Recurrence and Metastasis of Hepatocarcinoma Following Local Ablation
Status: Recruiting | Type: Observational
Sponsor: Yue Han (Other)
Responsible Party: Sponsor-Investigator, Yue Han, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Other Study IDs: HE-201708
Record Dates: First submitted 2017-11-12; First posted 2017-11-29 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Hepatocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation group 1: All treatments of patients after Local Ablation are prescribed by a physician on the basis of usual clinical practice.Patients who maybe receive Huaier Granule are as observation group 1
- Observation group 2: All treatments of patients after Local Ablation are prescribed by a physician on the basis of usual clinical practice.Patients who maybe not receive Huaier Granule are as observation group 2

SUMMARY:
To evaluate the efficacy and safety of Huaier Granule for Prevention of Recurrence and Metastasis of Hepatocarcinoma following Local Ablation

DETAILED DESCRIPTION:
A multicenter, prospective cohort study investigating Huaier Granule for Prevention of Recurrence and Metastasis of Hepatocarcinoma following Local Ablation，to evaluate the efficacy and safety

ELIGIBILITY:
Inclusion Criteria:

1. 18 years ≤ Age ≤ 75 years, both male and female
2. Patients are diagnosed with HCC via examination of tissues according to Guidelines for Diagnosis and Treatment of Hepatocellular Carcinoma (Version 2017) by NHFPC (National Health and Family Planning Commission of the People's Republic of China) and/or HCC imaging criteria of American Association for the Study of Liver Diseases (AASLD) for the diagnosis of HCC;
3. Radiographic testing shows cancer cells have been eliminated after four weeks of Local Ablation;Complete Response (CR): Dynamic contrast-enhanced CT scans and follow-up MR images show low-density area of Hepatocellular Carcinoma and no enhancement during the arterial phase of contrast-enhanced CT; also patients with 0.5-1 cm beyond the limits of the tumor margins (considered as safe surgical margins) are eligible;
4. According to contrast-enhanced CT and MRI, with solitary tumor smaller than 5 cm in diameter; with multiple tumors (no more than 3 masses), the largest dimension is less than 3 cm;
5. Patients are eligible if Hemoglobin (Hb) count ≥90g/L, platelets count (PLT) ≥60×109/L, absolute neutrophil count (ANC) count >1.0×109/L, prothrombin activity (PTA)>50%, serum creatinine is less than 1.5 times ULN (Upper Limit of Normal) and total bilirubin (TBIL) <51.3μmol/L (3 mg/dL);
6. ECOG score of 0-1;
7. Liver function is Child - Pugh grade A or B.
8. History of TACE for treatment of HCC is less than or equal to twice -
9. The patients are volunteered for the study, sign informed consent form and cooperate with Investigator to collect data.

Exclusion Criteria:

1. Radiographic testing shows cancer cells have not been eliminated after four weeks of Local Ablation;
2. The occurrence of embolism occurs in large blood vessels on liver, patients with extrahepatic metastatic of HCC or liver transplantation;
3. Patients who are about to receive or already received chemotherapy or molecular targeted therapy;
4. Patients who are about to receive TACE treatment for HCC;
5. Patients without previous treatment of Huaier granules.
6. History of diabetes;
7. HCC patients with uncontrollable ascites at the beginning of enrollment of the study or are very likely to have ascites during the next four weeks at the time of enrollment; patients with hepatic encephalopathy or upper gastrointestinal bleeding;
8. Patients have basic diseases including severe cardiopulmonary insufficiency, renal insufficiency, or severe mental illness;
9. Patients with other infectious disease (excluding viral hepatitis)
10. Patients who cannot take oral medication;
11. Conditions that are considered not suitable for this study investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatocellular Carcinoma patients after Local Ablation
Sampling Method: Non-Probability Sample
Enrollment: 828 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2024-08-26 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 96 weeks
  PFS was defined as the duration of time from start of treatment to time of disease progression.

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | 96 weeks
  RFS was defined as the duration of time from start of treatment to time of disease recurrence .
Time to recurrence (TTR) | Time from baseline to relapse (up to 96 weeks)
  TTR was defined as the time from shart of treatment to disease recurrence.
Overall Survival (OS) | Time from baseline to death (up to 96 weeks)
  OS was defined as the time from start to death from any cause or last patient last visit.
Change From Baseline in Quality of Life (QOL) | 24, 48, 72, 96 weeks
  Quality of Life (QOL) were measured using supplemental quality of life questions. Item score range（12 items）: 1 (worst symptom) to 5 (no symptom). Change: score at 96 weeks minus score at baseline.
Incidence rate of Adverse events (AE) | 96 weeks
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
severity of Adverse events (AE) | 96 weeks
  An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Han, Professor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (17):
- China (17):
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Shijiazhuang Fifth Hospital, Shijiazhuang, Hebei
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - the Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing You 'an Hospital, Capital Medical University, Beijing
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - Chinese PLA General Hospital, Beijing
  - Chongqing Cancer Hospital, Chongqing
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No